CLINICAL TRIAL: NCT00540943
Title: Phase I Study of Safety and Pharmacokinetics of Pazopanib in Combination With Cetuximab and Irinotecan in Patients With Colorectal Cancer
Brief Title: Study of Pazopanib, Irinotecan and Cetuximab in Combination to Treat 2nd Line Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG108925
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Colorectal
Keywords: cetuximab; irinotecan,; pazopanib,; Colorectal cancer,
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pazopanib; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): irinotecan and cetuximab in combination with pazopanib.
  Interventions: Drug: Pazopanib; Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: Pazopanib — Pazopanib is a potent, multi-targeted tyrosine kinase inhibitor of VEGFR-1, -2, -3, PDGFR-alpha and -beta and c-kit.
Drug: Cetuximab — Cetuximab will be supplied as a single-use 50 milliliter vial containing 100 micrograms of cetuximab as a sterile, preservative-free, injectable liquid at a concentration of 2 milligram per milliliter in phosphate.
  buffered saline
Drug: Irinotecan — Irinotecan hydrochloride trihydrate is an antineoplastic agent of the topoisomerase I inhibitor class.

SUMMARY:
Subjects will be entered into cohorts of 3 for the dose escalation phase so that the maximum tolerated dose can be determined. 18 additional patients will be recruited once the maximum tolerated dose (MTD) is determined for disease assessment.

ELIGIBILITY:
Inclusion criteria:

* Male or female at least 18 years of age.
* Willing and able to sign a written informed consent.
* Is either affiliated to or a beneficiary of a social security category
* Histologically or cytologically confirmed diagnosis of colorectal cancer. Subjects should have metastatic disease which is refractory or relapsed following prior treatment.
* Documented disease progression after prior treatment with 5-FU, oxaliplatin and irinotecan containing regimens.
* Complete recovery from surgical or radiotherapy procedures.
* Eastern Cooperative Oncology Group performance status of 0 or 1, or Karnofsky score ≥ 70%.
* Able to swallow and retain oral medications.
* Adequate bone marrow function (absolute neutrophil count greater than or equal to 1,500/mm3, platelet count greater than or equal to 100,000/mm3, hemoglobin levels greater than or equal to 10g/dL).
* Adequate renal function as determined by a creatinine clearance greater than 50 mL/minute calculated by the Cockcroft-Gault Formula. Measured creatinine clearance greater than or equal to 50 mL/minute by 24 hour urine collection will be acceptable in lieu of a calculated value.
* Urine Protein Creatinine (UPC) Ratio of ≤ 1 as assessed in a random or spot urine sample.
* Adequate hepatic function determined by total bilirubin within the normal range and aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT or SGPT) less than or equal to 2.5 times the upper limit of normal.
* Prothrombin time (PT), international normalized ratio (INR), and partial thromboplastin time (PTT) less than or equal to 1.2 times the ULN.
* A female subject is eligible to enter and participate in the study if she is:

  ·Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any woman who:
* Has had a hysterectomy, or
* Has had a bilateral oophorectomy (ovariectomy), or
* Has had a bilateral tubal ligation, or
* Is post-menopausal (demonstrate total cessation of menses for greater than or equal to 1 year).
* Childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following:
* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the subject's entry and is the sole sexual partner for that woman.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, throughout the clinical trial, and for at least 21 days after the last dose of investigational product.
* Double barrier contraception defined as condom with spermicidal jelly, foam, suppository, or film; OR diaphragm with spermicide; OR male condom and diaphragm.
* A male patient with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study.
* Predicted life expectancy of at least 12 weeks.
* Able to understand and comply with protocol requirements and instructions and intends to complete the study as planned.

Exclusion criteria:

* Has participated in any study using an investigational drug during the previous 28 days.
* Has had any major surgery, chemotherapy, investigational agent, or radiotherapy within the last 28 days and/or not recovered from prior therapy.
* Any history of grade III toxicity related to prior treatment with anti VEGF compound other than grade 3 hypertension subsequently controlled with antihypertensive agents.
* Has received prior treatment with pazopanib / investigational anti-angiogenic compounds or cetuximab. Prior treatment with Avastin is permitted. Known contraindications to the use of irinotecan and cetuximab.
* Unable to tolerate 180mg/m2 of irinotecan every two weeks during previous treatment.
* Is unable to discontinue prohibited medications, as stipulated in the protocol for 14 days prior to Visit 1 and for the duration of the study
* Has received Amiodarone for arrythmias within the last 6 months prior to Visit 1
* Has known allergy to penicillin.
* Women who are pregnant or lactating.
* Poorly controlled hypertension (systolic blood pressure [SBP] of 140 mmHg or higher, or diastolic blood pressure [DBP] of 90 mmHg or higher). Initiation or adjustment of blood pressure medication is permitted prior to study entry provided the subject has 2 consecutive blood pressure readings less than 140/90 mmHg, each separated by a minimum of 24 hours. These readings need to be collected prior to the first dose.
* Corrected QT (QTc) prolongation defined as a QTc interval greater than or equal to 480 msec and a prior history of cardiovascular disease, arrhythmias, or significant ECG abnormalities.
* Has Class III or IV heart failure as defined by the New York Heart Association functional classification system.
* Arterial thrombi, myocardial infarction, admission for unstable angina, uncontrolled or symptomatic arrhythmia, cardiac angioplasty, or stenting within the last 6 months.
* Any history of cerebrovascular accident (CVA), or pulmonary embolism within the last 6 months.
* History of untreated deep venous thrombosis (DVT) within the past 6 months (e.g. calf vein thrombosis). Note: Patients with recent DVT who have been treated with therapeutic anti-coagulant agents (excluding therapeutic warfarin) for at least 6 weeks are eligible.
* Current use of therapeutic warfarin. NOTE: Low molecular weight heparin and prophylactic low-dose warfarin (no more than 1mg per day) are permitted. PT/PTT and INR must be within 1.2 times the upper limit of normal.
* Known history of leptomeningeal or brain metastases. NOTE: Computed tomography or magnetic resonance imaging (MRI) scans are not required to rule out central nervous system metastases unless the subject is exhibiting neurologic signs or symptoms. If, however, CT or MRI scans are performed and document central nervous system disease, the subject is ineligible, regardless of whether neurologic signs or symptoms are present.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition (including laboratory abnormalities) that could interfere with subject safety or obtaining informed consent.
* History of mal-absorption syndrome, disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption, distribution, metabolism, or excretion of study drugs.
* History of any unresolved bowel obstruction or diarrhea.
* The subject has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, irinotecan, or cetuximab, unless enrolment is approved by the GSK Medical Monitor following discussion with the Investigator.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Is on any specifically prohibited medication or requires any of these medications during treatment with pazopanib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-07-13 (Actual); Primary Completion 2010-05-03 (Actual); Study Completion 2010-05-03 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of the maximum tolerated dose defined as a dose regimen where no more than 1 of 6 subjects experiences a dose limiting toxicity. | End of 2009

SECONDARY OUTCOMES:
pharmacokinetics disease assessment | 2010
Clearance of irinotecan (if data permit) and AUC, Cmax, tmax, and t1/2 of irinotecan and SN-38 after administration of irinotecan plus cetuximab. | 2010
AUC(0-24), Cmax, tmax, and t1/2 of pazopanib when administered with irinotecan and cetuximab | 2010
AUC(0-24), Cmax, and tmax of cetuximab when administered with irinotecan alone | 2010
AUC(0-24), Cmax, and tmax of cetuximab when administered with irinotecan plus pazopanib. | 2010
The ratio of SN-38 AUC(0-24) and irinotecan AUC(0-24) on Cycle 1 Day 1 and on Cycle 2 Day 1. | 2010
Objective response rate (complete response (CR) plus partial response (PR)) will be the primary measure of antitumor activity | 2010
Stable disease (SD) at 4 months | 4 months
Time to progression | 2010

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- France (2):
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Toulouse

REFERENCES:
- See also: Results for study VEG108925 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG108925?search=study&study_ids=VEG108925#rs